CLINICAL TRIAL: NCT03629184
Title: A Multicenter, Randomized, Double-Blind, Active (Oseltamivir)-Controlled Study to Assess the Safety, Pharmacokinetics, and Efficacy of Baloxavir Marboxil in Otherwise Healthy Pediatric Patients 1 to <12 Years of Age With Influenza-Like Symptoms
Brief Title: Study to Assess the Safety, Pharmacokinetics, and Efficacy of Baloxavir Marboxil in Healthy Pediatric Participants With Influenza-Like Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP40563; 2018-002169-21 (EudraCT Number)
Record Dates: First submitted 2018-08-10; First posted 2018-08-14 (Actual); Results first posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — baloxavir; Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Baloxavir Marboxil (Experimental): Participants will receive a single oral dose of baloxavir marboxil on Day 1 (based on body weight). Oseltamivir matching placebo will also be administered orally twice daily (BID) for 5 days.
  Interventions: Drug: Baloxavir Marboxil
- Oseltamivir (Active Comparator): Participants will receive oseltamivir orally BID for 5 days (based on body weight). Baloxavir marboxil matching placebo will also be administered orally on Day 1
  Interventions: Drug: Oseltamivir

INTERVENTIONS:
Drug: Baloxavir Marboxil — Baloxavir marboxil will be administered as oral suspension in a single dose on Day 1.
  Oseltamivir matching placebo will also be administered as oral suspension twice daily (BID) for 5 days.
  Arms: Baloxavir Marboxil
Drug: Oseltamivir — Oseltamivir will be administered as oral suspension BID for 5 days. Participants receiving oseltamivir will also receive baloxavir marboxil matching placebo as oral suspension, single dose on Day 1.
  Arms: Oseltamivir

SUMMARY:
This study will evaluate the safety, pharmacokinetics, and efficacy of baloxavir marboxil compared with oseltamivir in a single influenza episode in otherwise healthy pediatric participants (i.e., 1 to <12 years of age) with influenza-like symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Aged 1 to < 12 years at randomization (Day 1).
* Written informed consent/assent for study participation obtained from participant's parents or legal guardian, with assent as appropriate by the participant, depending on the patient's level of understanding
* Participant able to comply with study requirements, depending on the patient's level of understanding
* Participant with a diagnosis of influenza virus infection confirmed by the presence of all of the following:
* Fever ≥ 38 degree celsius (tympanic temperature) at screening
* At least one respiratory symptom (either cough or nasal congestion)
* The time interval between the onset of symptoms and screening is ≤ 48 hours

Exclusion Criteria:

* Severe symptoms of influenza virus infection requiring inpatient treatment
* Concurrent infections requiring systemic antiviral therapy at screening
* Require, in the opinion of the investigator, any of the prohibited medication during the study
* Previous treatment with peramivir, laninamivir, oseltamivir, zanamivir, or amantadine within 2 weeks prior to screening
* Immunization with a live/attenuated influenza vaccine in the 2 weeks prior to randomization
* Concomitant treatment with steroids or other immuno-suppressant therapy
* Known HIV infection or other immunosuppressive disorder
* Uncontrolled renal, vascular, neurologic, or metabolic disease (e.g., diabetes, thyroid disorders, adrenal disease), hepatitis, cirrhosis, or pulmonary disease or participants with known chronic renal failure.
* Active cancer at any site
* History of organ transplantation
* Known allergy to either study drug (i.e., baloxavir marboxil and oseltamivir) or to acetaminophen
* Females with child-bearing potential
* Participation in a clinical trial within 4 weeks or five half-lives of exposure to an investigational drug prior to screening, whichever is longer

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 173 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (37):
- United States (27):
  - Central Alabama Research; Pediatrics, Birmingham, Alabama
  - Harrisburg Family Medical Center, Harrisburg, Arkansas
  - The Children's Clinic of Jonesboro, P.A., Jonesboro, Arkansas
  - The Probe Medical Research, Los Angeles, California
  - Orange County Research Institute, Ontario, California
  - Khruz Biotechnology Research Institute, San Diego, California
  - Avanza Medical Research Center, Pensacola, Florida
  - Clinical Research Prime, Idaho Falls, Idaho
  - Cotton O'Neil Clinic; Stormont-Vail Hlth Care, Topeka, Kansas
  - Kentucky Pediatric Research Center, Bardstown, Kentucky
  - Spiegel, Craig, Bridgeton, Missouri
  - Meridian Clinical Research, Llc, Omaha, Nebraska
  - Machuca Family Medicine, Las Vegas, Nevada
  - OnSite Clinical Solutions LLC, Charlotte, North Carolina
  - Montgomery Medical Research /Frontier Clinical Research, Smithfield, North Carolina
  - Ohio Pediatric Research Association, Dayton, Ohio
  - Coastal Pediatric Research, Charleston, South Carolina
  - AFC Urgent Care- Cleveland, Cleveland, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Oak Cliff Research Company, LLC, Dallas, Texas
  - HD Research Corp, Houston, Texas
  - Mercury Clinical Research, Houston, Texas
  - Tekton Research, San Antonio, Texas
  - DM Clinical Research, Tomball, Texas
  - ClinPoint Trials, Waxahachie, Texas
  - FirstMed East (J Lewis Research), Salt Lake City, Utah
  - Advanced Clinical Research - Jordan Ridge Family Medicine, Salt Lake City, Utah
- ICIMED Instituto de Investigación en Ciencias Médicas, San José, Costa Rica
- Clalit Health Services- Pediatric Ambulatory Clinic; Pediatric Ambulatory Clinic, Petah Tikva, Israel
- Hospital San Jose; Centro de investigacion y transferencia en salud del Tec de Monterrey, Monterrey, N.L, Mexico
- Poland (4):
  - Wojewodzki Szpital Obserwacyjno-Zakazny; Oddział Pediatrii, Chorób Infekcyjnych i Hepatologii, Bydgoszcz
  - NZOZ Vitamed, Bydgoszcz
  - Prywatny Gabinet Lekarski, Dębica
  - NZLA Michalkowice Jarosz i partnerzy Spolka Lekarska, Siemianowice Śląskie
- MC Gepatolog, Samara, Russia
- Spain (2):
  - Complejo Hospitalario Universitario de Santiago (CHUS); Area Asistencial Integrada de Pediatría, Santiago de Compostela, LA Coruña
  - Hospital Universitario 12 de Octubre; Servicio de Pediatria, Madrid

REFERENCES:
- [Derived] Baker J, Block SL, Matharu B, Burleigh Macutkiewicz L, Wildum S, Dimonaco S, Collinson N, Clinch B, Piedra PA. Baloxavir Marboxil Single-dose Treatment in Influenza-infected Children: A Randomized, Double-blind, Active Controlled Phase 3 Safety and Efficacy Trial (miniSTONE-2). Pediatr Infect Dis J. 2020 Aug;39(8):700-705. doi: 10.1097/INF.0000000000002747. PMID 32516282

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Baloxavir Marboxil | Oseltamivir
Started | 115 | 58
Completed | 112 | 57
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Baloxavir Marboxil | Oseltamivir | Total
Number analyzed (Participants) | 115 | 58 | 173
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.10 (2.90) | 6.02 (3.20) | 6.08 (3.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 32 | 92
  Male | 55 | 26 | 81
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Black or African American | 6 | 5 | 11
  Native Hawaiian or other Pacific Islander | 0 | 1 | 1
  White | 98 | 51 | 149
  Multiple | 4 | 0 | 4
  Unknown | 5 | 1 | 6
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 52 | 27 | 79
  Not Hispanic or Latino | 63 | 31 | 94

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. A serious adverse event (SAE) is any significant hazard, contraindication, side effect that is fatal or life-threatening, requires hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability/ incapacity, is a congenital anomaly/ birth defect, is medically significant or requires intervention to prevent one or other of the outcomes listed above.
Time Frame: Up to Day 29
Measure: Number; unit: percentage of participants
Arm/Group | Baloxavir Marboxil | Oseltamivir
Number analyzed (Participants) | 115 | 58
percentage of participants
  Adverse Events (AEs) | 46.1 | 53.4
  Serious Adverse Events (SAEs) | 0 | 0

2. Secondary Outcome: Plasma Concentrations of Baloxavir Marboxil - Sparse PK Population
Description: Results provided by body-weight groups for participants in the Baloxavir Marboxil arm. Values below lower limit of quantification (0.5 ng/mL) are set to zero.
Time Frame: Days 1 (Post-Dose), 2, 4, 6 and 10
Population: The pharmacokinetic (PK) population consists of all participants that have at least one post-dose drug concentration measurement at a scheduled visit time point. Sparse PK population comprises all participants in the PK population who did not provide informed consent to intensive PK sampling
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 88
ng/mL
  5 - <10 kg (Day 1): number analyzed (Participants) | 1
  5 - <10 kg (Day 1) | 0.000 (NA) — Insufficient number of participants available to calculate the standard deviation
  5 - <10 kg (Day 2): number analyzed (Participants) | 1
  5 - <10 kg (Day 2) | 0.000 (NA) — Insufficient number of participants available to calculate the standard deviation
  5 - <10 kg (Day 4): number analyzed (Participants) | 0
  5 - <10 kg (Day 6): number analyzed (Participants) | 1
  5 - <10 kg (Day 6) | 0.000 (NA) — Insufficient number of participants available to calculate the standard deviation
  5 - <10 kg (Day 10): number analyzed (Participants) | 0
  10 - <15 kg (Day 1): number analyzed (Participants) | 16
  10 - <15 kg (Day 1) | 0.073 (0.2001)
  10 - <15 kg (Day 2): number analyzed (Participants) | 7
  10 - <15 kg (Day 2) | 0.000 (0.0000)
  10 - <15 kg (Day 4): number analyzed (Participants) | 9
  10 - <15 kg (Day 4) | 0.000 (0.0000)
  10 - <15 kg (Day 6): number analyzed (Participants) | 13
  10 - <15 kg (Day 6) | 0.000 (0.0000)
  10 - <15 kg (Day 10): number analyzed (Participants) | 3
  10 - <15 kg (Day 10) | 0.000 (0.0000)
  15 - <20 kg (Day 1): number analyzed (Participants) | 22
  15 - <20 kg (Day 1) | 0.090 (0.2386)
  15 - <20 kg (Day 2): number analyzed (Participants) | 13
  15 - <20 kg (Day 2) | 0.000 (0.0000)
  15 - <20 kg (Day 4): number analyzed (Participants) | 7
  15 - <20 kg (Day 4) | 0.000 (0.0000)
  15 - <20 kg (Day 6): number analyzed (Participants) | 17
  15 - <20 kg (Day 6) | 0.000 (0.0000)
  15 - <20 kg (Day 10): number analyzed (Participants) | 3
  15 - <20 kg (Day 10) | 0.000 (0.0000)
  >=20 kg (Day 1): number analyzed (Participants) | 58
  >=20 kg (Day 1) | 0.048 (0.1936)
  >=20 kg (Day 2): number analyzed (Participants) | 34
  >=20 kg (Day 2) | 0.000 (0.0000)
  >=20 kg (Day 4): number analyzed (Participants) | 25
  >=20 kg (Day 4) | 0.000 (0.0000)
  >=20 kg (Day 6): number analyzed (Participants) | 56
  >=20 kg (Day 6) | 0.000 (0.0000)
  >=20 kg (Day 10): number analyzed (Participants) | 6
  >=20 kg (Day 10) | 0.000 (0.0000)

3. Secondary Outcome: Plasma Concentrations of S-033447 - Sparse PK Population
Description: Results provided by body-weight groups for participants in the Baloxavir Marboxil arm.
Time Frame: Days 1 (Post-Dose), 2, 4, 6 and 10
Population: The PK population consists of all participants that have at least one post-dose drug concentration measurement at a scheduled visit time point. Sparse PK population comprises all participants in the PK population who did not provide informed consent to intensive PK sampling
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 88
ng/mL
  5 - <10 kg (Day 1): number analyzed (Participants) | 1
  5 - <10 kg (Day 1) | 45.700 (NA) — Insufficient number of participants available to calculate the standard deviation
  5 - <10 kg (Day 2): number analyzed (Participants) | 1
  5 - <10 kg (Day 2) | 45.800 (NA) — Insufficient number of participants available to calculate the standard deviation
  5 - <10 kg (Day 4): number analyzed (Participants) | 0
  5 - <10 kg (Day 6): number analyzed (Participants) | 1
  5 - <10 kg (Day 6) | 3.110 (NA) — Insufficient number of participants available to calculate the standard deviation
  5 - <10 kg (Day 10): number analyzed (Participants) | 0
  10 - <15 kg (Day 1): number analyzed (Participants) | 16
  10 - <15 kg (Day 1) | 49.084 (53.6689)
  10 - <15 kg (Day 2): number analyzed (Participants) | 7
  10 - <15 kg (Day 2) | 42.900 (16.5227)
  10 - <15 kg (Day 4): number analyzed (Participants) | 9
  10 - <15 kg (Day 4) | 9.233 (5.3879)
  10 - <15 kg (Day 6): number analyzed (Participants) | 13
  10 - <15 kg (Day 6) | 2.965 (1.6480)
  10 - <15 kg (Day 10): number analyzed (Participants) | 3
  10 - <15 kg (Day 10) | 0.367 (0.6351)
  15 - <20 kg (Day 1): number analyzed (Participants) | 22
  15 - <20 kg (Day 1) | 64.160 (73.6320)
  15 - <20 kg (Day 2): number analyzed (Participants) | 13
  15 - <20 kg (Day 2) | 67.729 (46.7346)
  15 - <20 kg (Day 4): number analyzed (Participants) | 7
  15 - <20 kg (Day 4) | 15.840 (10.8285)
  15 - <20 kg (Day 6): number analyzed (Participants) | 17
  15 - <20 kg (Day 6) | 4.829 (3.6562)
  15 - <20 kg (Day 10): number analyzed (Participants) | 3
  15 - <20 kg (Day 10) | 1.110 (1.9226)
  >=20 kg (Day 1): number analyzed (Participants) | 58
  >=20 kg (Day 1) | 29.899 (26.1558)
  >=20 kg (Day 2): number analyzed (Participants) | 34
  >=20 kg (Day 2) | 56.287 (40.4073)
  >=20 kg (Day 4): number analyzed (Participants) | 25
  >=20 kg (Day 4) | 18.674 (11.2179)
  >=20 kg (Day 6): number analyzed (Participants) | 56
  >=20 kg (Day 6) | 7.397 (5.0530)
  >=20 kg (Day 10): number analyzed (Participants) | 6
  >=20 kg (Day 10) | 3.953 (2.2536)

4. Secondary Outcome: Plasma Concentrations of Baloxavir Marboxil - Extensive PK Population
Description: as for outcome 2
Time Frame: Days 1 (Post-Dose), 2, 4, 6 and 10
Population: The PK population consists of all participants that have at least one post-dose drug concentration measurement at a scheduled visit time point. Extensive PK population comprises all participants in the PK population who provided informed consent to intensive PK sampling (additional time points for sample collection on Day 1)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 19
ng/mL
  Day 1, 0.5 - 2 hrs (5 - <10 kg): number analyzed (Participants) | 0
  Day 1, 4 hrs (5 - <10 kg): number analyzed (Participants) | 0
  Day 1, 6 hrs (5 - <10 kg): number analyzed (Participants) | 0
  Day 2 (5 - <10 kg): number analyzed (Participants) | 0
  Day 4 (5 - <10 kg ): number analyzed (Participants) | 0
  Day 6 (5 - <10 kg ): number analyzed (Participants) | 0
  Day 10 (5 - <10 kg): number analyzed (Participants) | 0
  Day 1, 0.5 - 2 hrs (10 - <15 kg): number analyzed (Participants) | 4
  Day 1, 0.5 - 2 hrs (10 - <15 kg) | 0.000 (0.0000)
  Day 1, 4 hrs (10 - <15 kg): number analyzed (Participants) | 2
  Day 1, 4 hrs (10 - <15 kg) | 0.000 (0.0000)
  Day 1, 6 hrs (10 - <15 kg): number analyzed (Participants) | 1
  Day 1, 6 hrs (10 - <15 kg) | 0.000 (NA) — Insufficient number of participants available to calculate the standard deviation
  Day 2 (10 - <15 kg): number analyzed (Participants) | 3
  Day 2 (10 - <15 kg) | 0.000 (0.0000)
  Day 4 (10 - <15 kg): number analyzed (Participants) | 1
  Day 4 (10 - <15 kg) | 0.000 (NA) — Insufficient number of participants available to calculate the standard deviation
  Day 6 (10 - <15 kg): number analyzed (Participants) | 3
  Day 6 (10 - <15 kg) | 0.000 (0.0000)
  Day 10 (10 - <15 kg ): number analyzed (Participants) | 1
  Day 10 (10 - <15 kg ) | 0.000 (NA) — Insufficient number of participants available to calculate the standard deviation
  Day 1, 0.5 - 2 hrs (15 - <20 kg): number analyzed (Participants) | 4
  Day 1, 0.5 - 2 hrs (15 - <20 kg) | 0.000 (0.0000)
  Day 1, 4 hrs (15 - <20 kg): number analyzed (Participants) | 1
  Day 1, 4 hrs (15 - <20 kg) | 0.000 (NA) — Insufficient number of participants available to calculate the standard deviation
  Day 1, 6 hrs (15 - <20 kg): number analyzed (Participants) | 1
  Day 1, 6 hrs (15 - <20 kg) | 0.000 (NA) — Insufficient number of participants available to calculate the standard deviation
  Day 2 (15 - <20 kg): number analyzed (Participants) | 2
  Day 2 (15 - <20 kg) | 0.000 (0.0000)
  Day 4 (15 - <20 kg): number analyzed (Participants) | 1
  Day 4 (15 - <20 kg) | 0.000 (NA) — Insufficient number of participants available to calculate the standard deviation
  Day 6 (15 - <20 kg): number analyzed (Participants) | 3
  Day 6 (15 - <20 kg) | 0.000 (0.0000)
  Day 10 (15 - <20 kg): number analyzed (Participants) | 0
  Day 1, 0.5 - 2 hrs (>=20 kg): number analyzed (Participants) | 10
  Day 1, 0.5 - 2 hrs (>=20 kg) | 0.051 (0.1600)
  Day 1, 4 hrs (>=20 kg): number analyzed (Participants) | 9
  Day 1, 4 hrs (>=20 kg) | 0.062 (0.1863)
  Day 1, 6 hrs ((>=20 kg): number analyzed (Participants) | 6
  Day 1, 6 hrs ((>=20 kg) | 0.000 (0.0000)
  Day 2 (>=20 kg): number analyzed (Participants) | 5
  Day 2 (>=20 kg) | 0.000 (0.0000)
  Day 4 (>=20 kg): number analyzed (Participants) | 4
  Day 4 (>=20 kg) | 0.000 (0.0000)
  Day 6 (>=20 kg): number analyzed (Participants) | 9
  Day 6 (>=20 kg) | 0.000 (0.0000)
  Day 10 (>=20 kg): number analyzed (Participants) | 0

5. Secondary Outcome: Plasma Concentrations of S-033447 - Extensive PK Population
Description: as for outcome 2
Time Frame: Days 1 (Post-Dose), 2, 4, 6 and 10
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 19
ng/mL
  Day 1, 0.5 - 2 hrs (5 - <10 kg): number analyzed (Participants) | 0
  Day 1, 4 hrs (5 - <10 kg): number analyzed (Participants) | 0
  Day 1, 6 hrs (5 - <10 kg): number analyzed (Participants) | 0
  Day 2 (5 - <10 kg): number analyzed (Participants) | 0
  Day 4 (5 - <10 kg ): number analyzed (Participants) | 0
  Day 6 (5 - <10 kg ): number analyzed (Participants) | 0
  Day 10 (5 - <10 kg): number analyzed (Participants) | 0
  Day 1, 0.5 - 2 hrs (10 - <15 kg): number analyzed (Participants) | 4
  Day 1, 0.5 - 2 hrs (10 - <15 kg) | 10.768 (14.7987)
  Day 1, 4 hrs (10 - <15 kg): number analyzed (Participants) | 2
  Day 1, 4 hrs (10 - <15 kg) | 49.500 (13.0108)
  Day 1, 6 hrs (10 - <15 kg): number analyzed (Participants) | 1
  Day 1, 6 hrs (10 - <15 kg) | 41.000 (NA) — Insufficient number of participants available to calculate the standard deviation
  Day 2 (10 - <15 kg): number analyzed (Participants) | 3
  Day 2 (10 - <15 kg) | 28.933 (14.7514)
  Day 4 (10 - <15 kg): number analyzed (Participants) | 1
  Day 4 (10 - <15 kg) | 2.230 (NA) — Insufficient number of participants available to calculate the standard deviation
  Day 6 (10 - <15 kg): number analyzed (Participants) | 3
  Day 6 (10 - <15 kg) | 3.131 (2.2828)
  Day 10 (10 - <15 kg ): number analyzed (Participants) | 1
  Day 10 (10 - <15 kg ) | 0.000 (NA) — Insufficient number of participants available to calculate the standard deviation
  Day 1, 0.5 - 2 hrs (15 - <20 kg): number analyzed (Participants) | 4
  Day 1, 0.5 - 2 hrs (15 - <20 kg) | 93.883 (152.5431)
  Day 1, 4 hrs (15 - <20 kg): number analyzed (Participants) | 1
  Day 1, 4 hrs (15 - <20 kg) | 72.900 (NA) — Insufficient number of participants available to calculate the standard deviation
  Day 1, 6 hrs (15 - <20 kg): number analyzed (Participants) | 1
  Day 1, 6 hrs (15 - <20 kg) | 80.300 (NA) — Insufficient number of participants available to calculate the standard deviation
  Day 2 (15 - <20 kg): number analyzed (Participants) | 2
  Day 2 (15 - <20 kg) | 42.640 (47.6024)
  Day 4 (15 - <20 kg): number analyzed (Participants) | 1
  Day 4 (15 - <20 kg) | 12.200 (NA) — Insufficient number of participants available to calculate the standard deviation
  Day 6 (15 - <20 kg): number analyzed (Participants) | 3
  Day 6 (15 - <20 kg) | 2.663 (1.5387)
  Day 10 (15 - <20 kg): number analyzed (Participants) | 0
  Day 1, 0.5 - 2 hrs (>=20 kg): number analyzed (Participants) | 10
  Day 1, 0.5 - 2 hrs (>=20 kg) | 19.923 (27.0980)
  Day 1, 4 hrs (>=20 kg): number analyzed (Participants) | 9
  Day 1, 4 hrs (>=20 kg) | 69.198 (55.7220)
  Day 1, 6 hrs ((>=20 kg): number analyzed (Participants) | 6
  Day 1, 6 hrs ((>=20 kg) | 65.527 (43.0799)
  Day 2 (>=20 kg): number analyzed (Participants) | 5
  Day 2 (>=20 kg) | 57.980 (37.8922)
  Day 4 (>=20 kg): number analyzed (Participants) | 4
  Day 4 (>=20 kg) | 21.775 (3.7968)
  Day 6 (>=20 kg): number analyzed (Participants) | 9
  Day 6 (>=20 kg) | 6.240 (3.3702)
  Day 10 (>=20 kg): number analyzed (Participants) | 0

6. Secondary Outcome: Time to Alleviation of Influenza Signs and Symptoms
Description: Time to alleviation of influenza signs and symptoms is defined as the length of time taken from the start of treatment to the point at which all of the following criteria are met and remain so for at least 21.5 hours:
  * A score of 0 (no problem) or 1 (minor problem) for cough and nasal symptoms (items 14 and 15 of the Canadian Acute Respiratory Illness and Flu Scale [CARIFS])
  * A "yes" response to the following question on the CARIFS: "Since the last assessment has the subject been able to return to day care/school, or resume his or her normal daily activity in the same way as performed prior to developing the flu?"
  * First return to afebrile state (tympanic temperature ≤37.2 degree Celsius [°C])
Time Frame: Up to Day 15
Population: Includes all participants with CARIFS Assessment who have had a laboratory confirmation of influenza infection (polymerase chain reaction [PCR] result) from any swab sample collected at baseline or during the study
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir Marboxil | Oseltamivir
Number analyzed (Participants) | 80 | 43
hours | 138.1 [116.6 to 163.2] | 150.0 [115.0 to 165.7]

7. Secondary Outcome: Duration of Fever
Description: Length of time taken by participants to return to afebrile state [tympanic temperature ≤ 37.2°C] and remaining so for at least 21.5 hours.
Time Frame: Up to Day 15
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir Marboxil | Oseltamivir
Number analyzed (Participants) | 80 | 43
hours | 41.2 [24.5 to 45.7] | 46.8 [30.0 to 53.5]

8. Secondary Outcome: Duration of Symptoms
Description: The clinical efficacy of baloxavir marboxil is evaluated by duration of symptoms i.e., alleviation of all symptoms as defined by a score of 0 [no problem] or 1 [minor problem] and remaining so for at least 21.5 hours, for all 18 symptoms specified in the CARIFS questionnaire.
Time Frame: Up to Day 15
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir Marboxil | Oseltamivir
Number analyzed (Participants) | 80 | 43
hours | 66.4 [43.7 to 76.4] | 67.9 [45.8 to 88.7]

9. Secondary Outcome: Time to Return to Normal Health and Activity
Description: Time to Return to Normal health and activity' is identified by a 'Yes' response to the following question on the CARIFS: "Since the last assessment has the patient been able to return to day care/school, or resume his or her normal daily activity in the same way as performed prior to developing the flu?"
Time Frame: Up to Day 15
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir Marboxil | Oseltamivir
Number analyzed (Participants) | 80 | 43
hours | 116.5 [94.9 to 138.0] | 111.6 [80.8 to 138.3]

10. Secondary Outcome: Frequency of Influenza-Related Complications
Description: Influenza related complications include death, hospitalization, radiologically confirmed pneumonia, bronchitis, sinusitis, otitis media, encephalitis/encephalopathy, febrile seizures, myositis.
Time Frame: Up to Day 29
Population: Includes all participants who have had a laboratory confirmation of influenza infection (polymerase chain reaction [PCR] result) from any swab sample collected at baseline or during the study
Measure: Number; unit: count of events
Arm/Group | Baloxavir Marboxil | Oseltamivir
Number analyzed (Participants) | 81 | 43
count of events
  Total | 6 | 4
  Death | 0 | 0
  Hospitalization | 0 | 0
  Sinusitis | 1 | 0
  Otitis Media | 3 | 3
  Pneumonia | 1 | 0
  Bronchitis | 1 | 0
  Encephalitis/Encephalopathy | 0 | 0
  Febrile Seizures | 0 | 1
  Myositis | 0 | 0

11. Secondary Outcome: Percentage of Participants With Influenza-Related Complications
Description: as for outcome 10
Time Frame: Up to Day 29
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Baloxavir Marboxil | Oseltamivir
Number analyzed (Participants) | 81 | 43
percentage of participants
  Total | 7.4 | 7.0
  Death | 0 | 0
  Hospitalization | 0 | 0
  Sinusitis | 1.2 | 0
  Otitis Media | 3.7 | 4.7
  Pneumonia | 1.2 | 0
  Bronchitis | 1.2 | 0
  Encephalitis/Encephalopathy | 0 | 0
  Febrile Seizures | 0 | 2.3
  Myositis | 0 | 0

12. Secondary Outcome: Percentage of Participants Requiring Antibiotics
Time Frame: Up to Day 29
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Baloxavir Marboxil | Oseltamivir
Number analyzed (Participants) | 81 | 43
percentage of participants
  Total | 4.9 | 4.7
  Bronchitis | 0 | 0
  Otitis Media | 2.5 | 4.7
  Pneumonia | 1.2 | 0
  Sinusitis | 1.2 | 0

13. Secondary Outcome: Time to Cessation of Viral Shedding by Virus Titer
Description: Time to cessation of viral shedding by virus titer is defined as the time, in hours, between the initiation of any study treatment and first time when the influenza virus titer is below the limit of detection.
Time Frame: Day 1 - Day 29
Population: Includes all participants with post-baseline Virology assessment and a positive virus titer on Day 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir Marboxil | Oseltamivir
Number analyzed (Participants) | 67 | 37
hours | 24.2 [23.5 to 24.6] | 75.8 [68.9 to 97.8]

14. Secondary Outcome: Time to Cessation of Viral Shedding by RT-PCR
Description: Time to cessation of viral shedding by RT-PCR, in hours, is defined as the time between the initiation of any study treatment and first time when the virus RNA by RT-PCR is below the limit of detection.
Time Frame: Day 1 - Day 29
Population: Includes all participants with post-baseline Virology assessment and a positive virus RNA by RT-PCR on Day 1. Participants whose virus RNA did not reach the limit by the last observation time point are treated as censored at that time point.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir Marboxil | Oseltamivir
Number analyzed (Participants) | 76 | 39
hours | 242.5 [235.8 to 262.8] | 238.9 [214.0 to 286.7]

15. Secondary Outcome: Change From Baseline in Influenza Virus Titer at Day 2, 4, 6, 10, 15, 29
Description: Influenza virus titer (log10TCID50/ML) is the quantity of influenza virus in a given volume within the samples obtained from nasal swabs. If influenza virus titer was less than the lower limit of quantification, the virus titer was imputed as 0.749 (log10TCID50/mL). A lower value indicates lower viral titer.
Time Frame: Baseline, Day 2, 3 (optional), 4, 6, 10, 15 (optional), 29
Population: Includes all participants with a positive virus titer on Day 1
Measure: Mean (Standard Deviation); unit: log10TCID50/ML
Arm/Group | Baloxavir Marboxil | Oseltamivir
Number analyzed (Participants) | 67 | 38
log10TCID50/ML
  Baseline | 4.43 (1.36) | 4.27 (1.48)
  Day 2: number analyzed (Participants) | 64 | 37
  Day 2 | -3.59 (1.34) | -1.79 (1.54)
  Day 3 (optional visit): number analyzed (Participants) | 3 | 2
  Day 3 (optional visit) | -2.83 (0.58) | -2.63 (0.88)
  Day 4: number analyzed (Participants) | 61 | 31
  Day 4 | -3.53 (1.38) | -3.27 (1.54)
  Day 6: number analyzed (Participants) | 63 | 35
  Day 6 | -3.55 (1.32) | -3.52 (1.50)
  Day 10: number analyzed (Participants) | 4 | 4
  Day 10 | -3.66 (1.40) | -3.50 (1.42)
  Day 15 (optional visit): number analyzed (Participants) | 4 | 4
  Day 15 (optional visit) | -3.75 (0.54) | -3.63 (1.45)
  Day 29: number analyzed (Participants) | 4 | 4
  Day 29 | -3.50 (1.43) | -3.75 (1.19)

16. Secondary Outcome: Change From Baseline in the Amount of Virus RNA (RT-PCR) at Day 2, 4, 6, 10, 15, 29
Description: If the amount of virus RNA was less than the lower limit of quantification, the amount of virus RNA was imputed as 2.18 for flu A and 2.93 for flu B (log10 virus particles/mL)
Time Frame: Baseline, Day 2, 3 (optional), 4, 6, 10, 15 (optional), 29
Population: Includes all participants with positive virus RNA by RT-PCR on Day 1
Measure: Mean (Standard Deviation); unit: log10 virus particles/mL
Arm/Group | Baloxavir Marboxil | Oseltamivir
Number analyzed (Participants) | 76 | 40
log10 virus particles/mL
  Baseline | 6.46 (1.50) | 6.86 (1.02)
  Day 2: number analyzed (Participants) | 70 | 39
  Day 2 | -1.74 (1.13) | -1.12 (1.12)
  Day 3 (optional): number analyzed (Participants) | 4 | 2
  Day 3 (optional) | -1.78 (1.50) | -2.21 (0.94)
  Day 4: number analyzed (Participants) | 61 | 30
  Day 4 | -2.40 (1.50) | -2.47 (1.35)
  Day 6: number analyzed (Participants) | 60 | 30
  Day 6 | -2.73 (1.78) | -3.32 (1.27)
  Day 10: number analyzed (Participants) | 35 | 15
  Day 10 | -3.55 (1.62) | -3.81 (1.19)
  Day 15 (optional): number analyzed (Participants) | 2 | 1
  Day 15 (optional) | -1.24 (3.06) | -4.44 (NA) — Insufficient number of participants available to calculate the standard deviation.
  Day 29: number analyzed (Participants) | 1 | 0
  Day 29 | 2.18 (NA) — Insufficient number of participants available to calculate the standard deviation. |

17. Secondary Outcome: Percentage of Participants With Positive Influenza Virus Titer at Day 2, 4, 6, 10
Time Frame: Baseline, Day 2, 3 (optional), 4, 6, 10
Population: Includes all participants with a positive virus titer on Day 1
Measure: Number; unit: percentage of participants
Arm/Group | Baloxavir Marboxil | Oseltamivir
Number analyzed (Participants) | 67 | 38
percentage of participants
  Baseline | 100 | 100
  Day 2: number analyzed (Participants) | 64 | 37
  Day 2 | 15.6 | 75.7
  Day 3 (optional): number analyzed (Participants) | 3 | 2
  Day 3 (optional) | 33.3 | 50.0
  Day 4: number analyzed (Participants) | 61 | 31
  Day 4 | 26.2 | 29.0
  Day 6: number analyzed (Participants) | 63 | 35
  Day 6 | 12.7 | 5.7
  Day 10: number analyzed (Participants) | 63 | 32
  Day 10 | 1.6 | 0

18. Secondary Outcome: Percentage of Participants Positive by RT-PCR at Day 2, 4, 6, 10, 15, 29
Time Frame: Day 2, 3 (optional), 4, 6, 10, 15 (optional), 29
Population: Includes all participants with positive virus RNA by RT-PCR on Day 1
Measure: Number; unit: percentage of participants
Arm/Group | Baloxavir Marboxil | Oseltamivir
Number analyzed (Participants) | 76 | 40
percentage of participants
  Baseline | 100 | 100
  Day 2: number analyzed (Participants) | 73 | 39
  Day 2 | 95.9 | 100
  Day 3 (optional): number analyzed (Participants) | 4 | 4
  Day 3 (optional) | 100 | 100
  Day 4: number analyzed (Participants) | 69 | 33
  Day 4 | 89.9 | 97.0
  Day 6: number analyzed (Participants) | 71 | 37
  Day 6 | 83.1 | 75.7
  Day 10: number analyzed (Participants) | 71 | 34
  Day 10 | 46.5 | 44.1
  Day 15 (optional): number analyzed (Participants) | 5 | 4
  Day 15 (optional) | 40.0 | 25.0
  Day 29: number analyzed (Participants) | 4 | 5
  Day 29 | 25.0 | 0

19. Secondary Outcome: Area Under the Curve in Virus Titer
Description: Area under the curve (AUC) in virus titer was calculated using the trapezoidal method.
Time Frame: Day 1 - Day 29
Population: Includes all participants with post-baseline Virology assessment and a positive virus titer on Day 1
Measure: Mean (Standard Deviation); unit: log₁₀[TCID₅₀/mL]*hours
Arm/Group | Baloxavir Marboxil | Oseltamivir
Number analyzed (Participants) | 67 | 37
log₁₀[TCID₅₀/mL]*hours | -863.81 (543.37) | -849.29 (684.43)

20. Secondary Outcome: Area Under the Curve in the Amount of Virus RNA (RT-PCR)
Description: AUC in virus RNA (RT-PCR) is defined as AUC of change from baseline in the amount of virus RNA (RT-PCR) from Day 1 to Day 10. AUC is calculated using the trapezoidal method similar to AUC in virus titer.
Time Frame: Day 1 - Day 10
Population: Includes all participants with positive virus RNA by RT-PCR on Day 1 and at least 1 post-baseline test.
Measure: Mean (Standard Deviation); unit: log₁₀ VPs/mL*hours
Arm/Group | Baloxavir Marboxil | Oseltamivir
Number analyzed (Participants) | 75 | 39
log₁₀ VPs/mL*hours | -381.53 (338.53) | -353.31 (304.01)

21. Secondary Outcome: Area Under the Concentration to Time Curve From Time 0 to Infinity (AUC0-inf) of Baloxavir Marboxil
Description: Dose groups correspond to body-weight groups. 2mg/kg dose was used for subjects <20 kgs and 40 mg dose was used for subjects >20 kgs.
Time Frame: Up to Day 10
Population: The PK population consists of all participants that have at least one post-dose drug concentration measurement at a scheduled visit time point
Measure: Mean (Standard Deviation); unit: ng.hr/mL
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 95
ng.hr/mL
  Non-Asian - 2 mg/kg: number analyzed (Participants) | 36
  Non-Asian - 2 mg/kg | NA (NA) — Not estimable as Baloxavir marboxil is a prodrug which is rapidly metabolised into baloxavir. The concentrations are not measurable and do not allow to derive any PK parameters.
  Asian - 40 mg: number analyzed (Participants) | 1
  Asian - 40 mg | NA (NA) — Not estimable as Baloxavir marboxil is a prodrug which is rapidly metabolised into baloxavir. The concentrations are not measurable and do not allow to derive any PK parameters.
  Non-Asian - 40 mg: number analyzed (Participants) | 58
  Non-Asian - 40 mg | NA (NA) — Not estimable as Baloxavir marboxil is a prodrug which is rapidly metabolised into baloxavir. The concentrations are not measurable and do not allow to derive any PK parameters.

22. Secondary Outcome: Area Under the Concentration to Time Curve From Time 0 to Infinity (AUC0-inf) of S-033447.
Description: as for outcome 21
Time Frame: Up to Day 10
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ng.hr/mL
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 95
ng.hr/mL
  Non-Asian - 2 mg/kg: number analyzed (Participants) | 36
  Non-Asian - 2 mg/kg | 4050 (2080)
  Asian - 40 mg: number analyzed (Participants) | 1
  Asian - 40 mg | 6600 (NA) — Not estimable due to low number of events
  Non-Asian - 40 mg: number analyzed (Participants) | 58
  Non-Asian - 40 mg | 4390 (2080)

23. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Baloxavir Marboxil
Description: as for outcome 21
Time Frame: Up to Day 10
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 95
ng/mL
  Non-Asian - 2 mg/kg: number analyzed (Participants) | 36
  Non-Asian - 2 mg/kg | NA (NA) — Not estimable as Baloxavir marboxil is a prodrug which is rapidly metabolised into baloxavir. The concentrations are not measurable and do not allow to derive any PK parameters.
  Asian - 40 mg: number analyzed (Participants) | 1
  Asian - 40 mg | NA (NA) — Not estimable as Baloxavir marboxil is a prodrug which is rapidly metabolised into baloxavir. The concentrations are not measurable and do not allow to derive any PK parameters.
  Non-Asian - 40 mg: number analyzed (Participants) | 58
  Non-Asian - 40 mg | NA (NA) — Not estimable as Baloxavir marboxil is a prodrug which is rapidly metabolised into baloxavir. The concentrations are not measurable and do not allow to derive any PK parameters.

24. Secondary Outcome: Maximum Plasma Concentration (Cmax) of S-033447
Description: as for outcome 21
Time Frame: Up to Day 10
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 95
ng/mL
  Non-Asian - 2 mg/kg: number analyzed (Participants) | 36
  Non-Asian - 2 mg/kg | 109 (55.3)
  Asian - 40 mg: number analyzed (Participants) | 1
  Asian - 40 mg | 110 (NA) — Not estimable due to low number of events.
  Non-Asian - 40 mg: number analyzed (Participants) | 58
  Non-Asian - 40 mg | 83.2 (36.5)

25. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Baloxavir Marboxil
Description: as for outcome 21
Time Frame: Up to Day 10
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 95
hours
  Non-Asian - 2 mg/kg: number analyzed (Participants) | 36
  Non-Asian - 2 mg/kg | NA (NA) — Not estimable as Baloxavir marboxil is a prodrug which is rapidly metabolised into baloxavir. The concentrations are not measurable and do not allow to derive any PK parameters.
  Asian - 40 mg: number analyzed (Participants) | 1
  Asian - 40 mg | NA (NA) — Not estimable as Baloxavir marboxil is a prodrug which is rapidly metabolised into baloxavir. The concentrations are not measurable and do not allow to derive any PK parameters.
  Non-Asian - 40 mg: number analyzed (Participants) | 58
  Non-Asian - 40 mg | NA (NA) — Not estimable as Baloxavir marboxil is a prodrug which is rapidly metabolised into baloxavir. The concentrations are not measurable and do not allow to derive any PK parameters.

26. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of S-033447
Description: as for outcome 21
Time Frame: Up to Day 10
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 95
hours
  Non-Asian - 2 mg/kg: number analyzed (Participants) | 36
  Non-Asian - 2 mg/kg | 4.12 (2.07)
  Asian - 40 mg: number analyzed (Participants) | 1
  Asian - 40 mg | 5.50 (NA) — Not estimable due to low number of events
  Non-Asian - 40 mg: number analyzed (Participants) | 58
  Non-Asian - 40 mg | 5.55 (3.79)

27. Secondary Outcome: Plasma Concentrations of Baloxavir Marboxil by Dosage
Description: as for outcome 21
Time Frame: 24, 72, 96 and 240 hours post-dose
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 95
ng/mL
  24 - Non-Asian - 2 mg/kg: number analyzed (Participants) | 36
  24 - Non-Asian - 2 mg/kg | NA (NA) — Not estimable as Baloxavir marboxil is a prodrug which is rapidly metabolised into baloxavir. The concentrations are not measurable and do not allow to derive any PK parameters.
  24 - Asian - 40 mg: number analyzed (Participants) | 1
  24 - Asian - 40 mg | NA (NA) — Not estimable as Baloxavir marboxil is a prodrug which is rapidly metabolised into baloxavir. The concentrations are not measurable and do not allow to derive any PK parameters.
  24 - Non-Asian - 40 mg: number analyzed (Participants) | 58
  24 - Non-Asian - 40 mg | NA (NA) — Not estimable as Baloxavir marboxil is a prodrug which is rapidly metabolised into baloxavir. The concentrations are not measurable and do not allow to derive any PK parameters.
  72 - Non-Asian - 2 mg/kg: number analyzed (Participants) | 36
  72 - Non-Asian - 2 mg/kg | NA (NA) — Not estimable as Baloxavir marboxil is a prodrug which is rapidly metabolised into baloxavir. The concentrations are not measurable and do not allow to derive any PK parameters.
  72 - Asian - 40 mg: number analyzed (Participants) | 1
  72 - Asian - 40 mg | NA (NA) — Not estimable as Baloxavir marboxil is a prodrug which is rapidly metabolised into baloxavir. The concentrations are not measurable and do not allow to derive any PK parameters.
  72 - Non-Asian - 40 mg: number analyzed (Participants) | 58
  72 - Non-Asian - 40 mg | NA (NA) — Not estimable as Baloxavir marboxil is a prodrug which is rapidly metabolised into baloxavir. The concentrations are not measurable and do not allow to derive any PK parameters.
  96 - Non-Asian - 2 mg/kg: number analyzed (Participants) | 36
  96 - Non-Asian - 2 mg/kg | NA (NA) — Not estimable as Baloxavir marboxil is a prodrug which is rapidly metabolised into baloxavir. The concentrations are not measurable and do not allow to derive any PK parameters.
  96 - Asian - 40 mg: number analyzed (Participants) | 1
  96 - Asian - 40 mg | NA (NA) — Not estimable as Baloxavir marboxil is a prodrug which is rapidly metabolised into baloxavir. The concentrations are not measurable and do not allow to derive any PK parameters.
  96 - Non-Asian - 40 mg: number analyzed (Participants) | 58
  96 - Non-Asian - 40 mg | NA (NA) — Not estimable as Baloxavir marboxil is a prodrug which is rapidly metabolised into baloxavir. The concentrations are not measurable and do not allow to derive any PK parameters.
  240 - Non-Asian - 2 mg/kg: number analyzed (Participants) | 36
  240 - Non-Asian - 2 mg/kg | NA (NA) — Not estimable as Baloxavir marboxil is a prodrug which is rapidly metabolised into baloxavir. The concentrations are not measurable and do not allow to derive any PK parameters.
  240 - Asian - 40 mg: number analyzed (Participants) | 1
  240 - Asian - 40 mg | NA (NA) — Not estimable as Baloxavir marboxil is a prodrug which is rapidly metabolised into baloxavir. The concentrations are not measurable and do not allow to derive any PK parameters.
  240 - Non-Asian - 40 mg: number analyzed (Participants) | 58
  240 - Non-Asian - 40 mg | NA (NA) — Not estimable as Baloxavir marboxil is a prodrug which is rapidly metabolised into baloxavir. The concentrations are not measurable and do not allow to derive any PK parameters.

28. Secondary Outcome: Plasma Concentrations of S-033447 by Dosage
Description: as for outcome 21
Time Frame: 24, 72, 96 and 240 hours post-dose
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 95
ng/mL
  24 - Non-Asian - 2 mg/kg: number analyzed (Participants) | 36
  24 - Non-Asian - 2 mg/kg | 55.7 (28.1)
  24 - Asian - 40 mg: number analyzed (Participants) | 1
  24 - Asian - 40 mg | 75.2 (NA) — Not estimable due to low number of events
  24 - Non-Asian - 40 mg: number analyzed (Participants) | 58
  24 - Non-Asian - 40 mg | 53.2 (22.4)
  72 - Non-Asian - 2 mg/kg: number analyzed (Participants) | 36
  72 - Non-Asian - 2 mg/kg | 13.2 (7.15)
  72 - Asian - 40 mg: number analyzed (Participants) | 1
  72 - Asian - 40 mg | 28.9 (NA) — Not estimable due to low number of events
  72 - Non-Asian - 40 mg: number analyzed (Participants) | 58
  72 - Non-Asian - 40 mg | 17.90 (8.910)
  96 - Non-Asian - 2 mg/kg: number analyzed (Participants) | 36
  96 - Non-Asian - 2 mg/kg | 7.61 (4.400)
  96 - Asian - 40 mg: number analyzed (Participants) | 1
  96 - Asian - 40 mg | 19.0 (NA) — Not estimable due to low number of events
  96 - Non-Asian - 40 mg: number analyzed (Participants) | 58
  96 - Non-Asian - 40 mg | 11.3 (6.160)
  240 - Non-Asian - 2 mg/kg: number analyzed (Participants) | 36
  240 - Non-Asian - 2 mg/kg | 0.989 (0.887)
  240 - Asian - 40 mg: number analyzed (Participants) | 1
  240 - Asian - 40 mg | 3.31 (NA) — Not estimable due to low number of events
  240 - Non-Asian - 40 mg: number analyzed (Participants) | 58
  240 - Non-Asian - 40 mg | 1.85 (1.400)

ADVERSE EVENTS:
Time Frame: From baseline (Day 1) until 28 days after the last dose of study drug (29 days)
Arm/Group | Baloxavir Marboxil | Oseltamivir
All-Cause Mortality (participants affected / at risk) | 0/115 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/115 | 0/58
Other Adverse Events (participants affected / at risk) | 15/115 | 13/58
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baloxavir Marboxil (N=115) | Oseltamivir (N=58)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (7) | 9 (10)
Otitis Media (Infections and infestations) | 3 (3) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-06-29): https://cdn.clinicaltrials.gov/large-docs/84/NCT03629184/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-24): https://cdn.clinicaltrials.gov/large-docs/84/NCT03629184/SAP_001.pdf